CLINICAL TRIAL: NCT05054192
Title: Evaluation of Test-retest Reliability, Concurrent Validity and Minimal Detectable Change of the Modified Four Square Step Test in Individuals With Primary Total Hip Arthroplasty.
Brief Title: Reliability and Validity of Modified Four Square Step Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2021/414
Record Dates: First submitted 2021-09-10; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Total Hip Arthroplasty
Keywords: Postural Balance; Total Hip Arthroplasty; Falling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional improvements are reached in patients with primary total hip arthroplasty compared to the pre-operative term however some problems as continued range of motion limitations, loss of joint proprioception sensation, and resulting balance and gait disorders may result in failure of the Four Square Step Test. Therefore, the need for the apply of the Modified Four Square Step Test in individuals with primary THA is necessary. The aim of this study is to evaluate the test-retest reliability, concurrent validity and minimal detectable change of the Modified Four Square Step Test in individuals with primary total hip arthroplasty.

DETAILED DESCRIPTION:
Roos et al. improved the Modified Four-Square Step Test to complete the test by stroke patients and not to fall due to practices of the test while performing the test. The Modified Four Square Step Test variates from the The Four Square Step Test is that the person is not asked to look ahead during the test, and instead of using a cane, tapes are used to prevent people from losing their balance by tripping over the obstacle. Thus, although the height of the obstacle is reduced, the boundaries of the obstacle are preserved.

Functional improvements are reached in patients with primary total hip arthroplasty compared to the pre-operative term however some problems as continued range of motion limitations, loss of joint proprioception sensation, and resulting balance and gait disorders may result in failure of the Four Square Step Test. Therefore, the need for the apply of the Modified Four Square Step Test in individuals with primary THA is necessary. The aim of this study is to evaluate the test-retest reliability, concurrent validity and minimal detectable change of the Modified Four Square Step Test in individuals with primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-85.
* Having undergone primary total hip arthroplasty at least ≥6 months ago.

Exclusion Criteria:

* Having severe cardiovascular or lung disease
* Having severe dementia or communication difficulties
* Having a musculoskeletal or neurological problem that may affect participation in balance tests
* Having an uncorrectable visual impairment
* Having a body mass index of more than 40 kg/m2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, the participants will consist of individuals who have previously undergone primary total hip arthroplasty in Afyonkarahisar Health Sciences University Health Practice and Research Center Orthopedics and Traumatology Polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance | 6 minutes
  Dynamic balance is the ability of an object to balance while in motion or switching between positions. Dynamic balance will be evaluated with the modified four square step test. The duration as second will be recorded.

SECONDARY OUTCOMES:
Dynamic Balance | 4 minutes
  Dynamic balance will be evaluated with the timed and go test and the test completion time will be recorded in seconds.
Dynamic Balance | 25 minutes
  Dynamic balance will be evaluated with the Berg Balance Test. The scores from the test will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — Afyonkarahisar Health Science University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)